CLINICAL TRIAL: NCT00269802
Title: Multicenter Study Comparing the Efficacy and Safety of OROS (Methylphenidate HCl), Ritalin, and Placebo in Children With ADHD
Brief Title: A Multicenter Study Comparing the Efficacy and Safety of OROS Methylphenidate HCl, Ritalin (Methylphenidate HCl) and Placebo in Children With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005995
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Attention Deficit Hyperactivity Disorder; OROS®; Ritalin®; children; methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

ARMS (3):
- 001 (Experimental): OROS methylphenidate HCl
  Interventions: Drug: OROS methylphenidate HCl
- 002 (Active Comparator): Ritalin
  Interventions: Drug: Ritalin
- 003 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OROS methylphenidate HCl
  Arms: 001
Drug: Ritalin
  Arms: 002
Drug: Placebo
  Arms: 003

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of OROSÂ® Methylphenidate HCl as compared with placebo and standard immediate-release RitalinÂ® (taken three time per day) for the treatment of Attention Deficit Hyperactivity Disorder in children. Both OROSÂ® Methylphenidate HCl and RitalinÂ® contain the central nervous system stimulant, methylphenidate HCl.

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity Disorder (ADHD) represents the most common neurobehavioral disorder in children, affecting 3% to 5% of the school-age population. Behavioral pediatricians, child psychiatrists, and child neurologists indicate that referrals for ADHD may constitute up to 50% of their practices. This is a multicenter, double-blind, double-dummy, randomized, placebo-controlled, active-controlled, three-treatment, parallel group study to evaluate the efficacy and safety of OROS® (methylphenidate HCl) with standard immediate-release Ritalin® (three times a day), and placebo, in children with ADHD. Patients are assigned to one of three treatments, depending upon their prestudy titrated therapeutic dose and regimen, and are treated for 28 days. Patients will be given OROS® (methylphenidate HCl), 18, 36 or 54 milligrams once daily, or Ritalin® 5, 10, or 15 milligrams (encapsulated/single capsule) three times a day, or placebo. Efficacy is evaluated in the community setting by teachers, parents and investigators using standardized attention and behavior scales and other assessments. The primary measure of effectiveness is the teacher's rating on study Day 27 on the IOWA Conners Inattention/Overactivity subscale. Additional measures of effectiveness include the IOWA Conners Oppositional/Defiance subscale ratings, peer interaction and other behavioral ratings, SNAP-IV ratings, global assessments of efficacy, investigator Clinical Global Impression (CGI), home situation and the parent satisfaction questionnaire. Safety evaluations include the incidence of adverse events, physical examinations, clinical laboratory tests, vital signs, sleep quality, appetite, and the presence/severity of tics (hard-to-control, repeated twitching of any parts of the body or hard-to-control repeating of sounds or words). Patients will be given orally for 28 days: OROS® (methylphenidate HCl), 1, 2, or 3 of the 18 milligram tablets once daily, or Ritalin® 5, 10, or 15 milligrams (encapsulated/single capsule) three times daily, or placebo

ELIGIBILITY:
Inclusion Criteria:

* Patients who have successfully completed the ALZA screening protocol C-98-011 within the past six months
* taking or have taken in the past 5 - 20 mg of immediate-release methylphenidate (Ritalin®) at least twice a day, 20 - 60 mg of sustained-release methylphenidate (Ritalin-SR®) per day, or a combination of immediate-release and sustained-release methylphenidate up to a daily dose not exceeding 60 mg, or have successfully completed ALZA Protocol C-98-007
* agreeing to take only the supplied study drug as treatment for ADHD during the four-week treatment phase of the study
* who are able to comply with the study visit schedule and whose parent(s) and teacher are willing and able to complete the protocol-specified assessments
* having normal urinalysis, hematological and blood chemistry values or, if values are outside the normal range, they are determined to be not clinically significant by the investigator

Exclusion Criteria:

* Patients who have clinically significant gastrointestinal problems, including narrowing of the gastrointestinal tract
* having glaucoma, an ongoing seizure disorder, a psychotic disorder, clinical depression (and are suicidal or require immediate treatment for depression), or a diagnosis of Tourette's syndrome
* having a known allergy to methylphenidate or currently having significant adverse experiences from methylphenidate
* having a mean of two blood pressure measurements (systolic or diastolic) equal to or greater than the 95th percentile for age, sex, and height at screening
* if female, have begun menstruation

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Study Completion 1999-02 (Actual)

PRIMARY OUTCOMES:
IOWA Conners Rating Scale (Inattention/Overactivity subscale) rating by the teacher on Day 27.

SECONDARY OUTCOMES:
Teacher's IOWA Conners (Inattention/Overactivity and Oppositional Defiance subscales) rating on Days 1, 6, 13, 20, and 27; Incidence of adverse events; Changes in physical exams, laboratory tests, vital signs, sleep quality, appetite, and tics

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA

REFERENCES:
- [Result] Wolraich ML, Greenhill LL, Pelham W, Swanson J, Wilens T, Palumbo D, Atkins M, McBurnett K, Bukstein O, August G. Randomized, controlled trial of oros methylphenidate once a day in children with attention-deficit/hyperactivity disorder. Pediatrics. 2001 Oct;108(4):883-92. doi: 10.1542/peds.108.4.883. PMID 11581440